CLINICAL TRIAL: NCT04344938
Title: Covid 19 Pandemic. Emerging Legal and Ehical Disputes Over Patient Confidentiality
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Collaborators: Doaa M.EL Shehaby (Unknown)
Responsible Party: Principal Investigator, Noha Esmael Ebrahem, lecturer of forensic medicine and clinical toxicology, Assiut University
Other Study IDs: 2020A10
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Covid 19 Pandemic From Ethical View

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- medical personel
  Interventions: Other: questionnair about Emerging Legal and Ehical Disputes Over Patient Confidentiality
- non medical personel
  Interventions: Other: questionnair about Emerging Legal and Ehical Disputes Over Patient Confidentiality

INTERVENTIONS:
Other: questionnair about Emerging Legal and Ehical Disputes Over Patient Confidentiality — Many critical ethical questions arise in pandemic covid 19planning, preparedness and response. These include: Who will get priority access to medications, vaccines and intensive care unit beds, given the potential shortage of these essential resources? In the face of a pandemic, what obligations do health-care workers have to work notwithstanding risks to their own health and the health of their families? How can surveillance, isolation, quarantine and social-distancing measures be undertaken in a way that respects ethical norms? What obligations do countries have to one another with respect to pandemic covid 19 planning and response efforts?

SUMMARY:
Many critical ethical questions arise in pandemic covid 19planning, preparedness and response. These include: Who will get priority access to medications, vaccines and intensive care unit beds, given the potential shortage of these essential resources? In the face of a pandemic, what obligations do health-care workers have to work not withstanding risks to their own health and the health of their families? How can surveillance, isolation, quarantine and social-distancing measures be undertaken in a way that respects ethical norms? What obligations do countries have to one another with respect to pandemic covid 19 planning and response efforts?

ELIGIBILITY:
Inclusion Criteria:

* adult aged 18 years to 60 years
* medical personel graduated from egyptian faculty of medicine.
* non medical personel live in egypt

Exclusion Criteria:

* personel less than 18 years old .
* medical personel not graduated from egyptian faculty of medicine.
* non medical personel live outside egypt

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: medical and non medical personel
Sampling Method: Probability Sample
Enrollment: 874 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate the ethical requirement of controlled disrupts of patients In case of infectious disease pandemic | 2 months
  questionaire done to To keep the general preventive measure in the community